CLINICAL TRIAL: NCT07129681
Title: A Comparison of the Outcomes Following Intra-articular Dextrose 5% Injection Versus Arthrocentesis in Patients With Anterior Disc Displacement With Reduction of the Temporomandibular Joint.
Brief Title: a Comparison of the Outcomes Following Intra-articular Dextrose 5% Injection Versus Arthrocentesis in Patients With Anterior Disc Displacement With Reduction of the Tomporomandibular Joint
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sandy maged habib ibrahim, sandy Maged Habib Ibrahim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dextrose 5% injection in TMJ
Record Dates: First submitted 2025-07-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: TMJ Disc Disorder
Keywords: TMJ; Disc displacement with reduction; Dextrose 5%; Arthrocentesis
MeSH Terms: interventions — Arthrocentesis; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 patients with anterior disc displacement with reduction (Active Comparator)
  Interventions: Other: dextrose 5%
- Group 2 patients with anterior disc displacement of reduction (Experimental)
  Interventions: Other: Arthrocentesis/Saline

INTERVENTIONS:
Other: dextrose 5% — Dextrose, is an osmotic proliferant which acts by dehydrating the cells at the injection site which utlimately leads to release of cellular fragments that act as chemo attractants and start the inflammatory cascade leading todeposition of collagen
  Arms: Group 1 patients with anterior disc displacement with reduction
Other: Arthrocentesis/Saline — Arthrocentesis , a highly successful, simple and minimally invasive procedure is a safe and simple method for treatment of anterior disc displacement with reduction of TMJ both in short term and long term follow up period, where it is a procedure of removing damaged tissues &inflammatory mediators.it can be the treatment modality for the for control group
  Arms: Group 2 patients with anterior disc displacement of reduction

SUMMARY:
The Aim of this study is to evaluate the efficacy of intra-articular Dextrose injection with

concentration 5% in superior joint space of TMJ in comparison to arthrocentesis in patients with

anterior disc displacement with reduction of TMJ who did not respond favorably to conservative

treatment and to compare and infer which among the two procedures is more satisfactory,

whether dextrose 5% injection or Arthrocentesis.

DETAILED DESCRIPTION:
The Aim of this study is to evaluate the efficacy of intra-articular Dextrose injection with

concentration 5% in superior joint space of TMJ in comparison to arthrocentesis in patients with

anterior disc displacement with reduction of TMJ who did not respond favorably to conservative

treatment and to compare and infer which among the two procedures is more satisfactory,

whether dextrose 5% injection or Arthrocentesis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

-Patients diagnosed with anterior disc displacement with reduction of TMJ with pain,limited mouth opening and

painful clicking who underwent conservative therapy with physiotherapy but failed to receive any relief after 3

months of conservative therapy.

* Age ranges from 18 to 50 years.
* Patients with adequate follow up duration for outcome assessment.

Exclusion Criteria:

* Patients having pain or reduced mouth opening due to fracture of the condyle.
* patients having any degenerative changes in the TMJ.
* patients having other systemic diseases such as polyarthritis.
* patients having any neurological disorders.
* Pregnant and lactating women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Severity Measured by Numerical Rating Scale (NRS) | Measured at baseline, 3 days and 3 months after injection
  Primary Outcome Measure:
  1. Change in Pain Severity Measured by Numerical Rating Scale (NRS)
  Pain severity will be assessed using the Numerical Rating Scale (NRS) (0-10), where 0 = no pain and 10 = severe
  pain. Participants will report their pain levels at each time point. The mean change in NRS scores from baseline will be
  calculated and analyzed . Data Aggregation: Mean change in NRS score

SECONDARY OUTCOMES:
Change in Maximal Interincisal Opening (MIO) Measured in Millimeters | Measured at baseline, 3 days and 3 months after injection
  Maximal interincisal opening (MIO) will be measured using a sterilllized metal scale or a digital caliper, with values recorded in millimeters (mm).
  The mean change in MIO from baseline will be reported . Data Aggregation: Mean change in MIO (mm) with standard
  deviation (SD).

OTHER OUTCOMES:
Presence or Absence of Joint Clicking (Binary Outcome) | Measured at baseline, 3 days and 3 months after injection
  Joint clicking will be assessed as a binary outcome (Yes/No) based on clinical examination and patient-reported
  symptoms. The percentage of participants with joint clicking at each time point will be reported.
  Data Aggregation: Percentage of participants with joint clicking at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Mohamed Talaat, Cairo assistant professor, PHD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karadayi U, Gursoytrak B. Randomised controlled trial of arthrocentesis with or without PRF for internal derangement of the TMJ. J Craniomaxillofac Surg. 2021 May;49(5):362-367. doi: 10.1016/j.jcms.2021.01.018. Epub 2021 Feb 5. PMID 33581954
- [Background] Young AL. Internal derangements of the temporomandibular joint: A review of the anatomy, diagnosis, and management. J Indian Prosthodont Soc. 2015 Jan-Mar;15(1):2-7. doi: 10.4103/0972-4052.156998. PMID 26929478
- [Background] Maniquis-Smigel L, Dean Reeves K, Jeffrey Rosen H, Lyftogt J, Graham-Coleman C, Cheng AL, Rabago D. Short Term Analgesic Effects of 5% Dextrose Epidural Injections for Chronic Low Back Pain: A Randomized Controlled Trial. Anesth Pain Med. 2016 Dec 6;7(1):e42550. doi: 10.5812/aapm.42550. eCollection 2017 Feb. PMID 28920043
- [Background] Rabago D, Mundt M, Zgierska A, Grettie J. Hypertonic dextrose injection (prolotherapy) for knee osteoarthritis: Long term outcomes. Complement Ther Med. 2015 Jun;23(3):388-95. doi: 10.1016/j.ctim.2015.04.003. Epub 2015 Apr 8. PMID 26051574
- [Background] Fouda AA. Change of site of intra-articular injection of hypertonic dextrose resulted in different effects of treatment. Br J Oral Maxillofac Surg. 2018 Oct;56(8):715-718. doi: 10.1016/j.bjoms.2018.07.022. Epub 2018 Aug 11. PMID 30107954
- [Background] Singh SU, Prasad RB, Punga R, Datta R, Singh N. A comparison of the outcomes following intra-articular steroid injection alone or arthrocentesis alone in the management of internal derangement of the temporomandibular joint. Natl J Maxillofac Surg. 2022 Aug;13(Suppl 1):S80-S84. doi: 10.4103/njms.njms_291_21. Epub 2022 Aug 20. PMID 36393924
- [Background] Li TY, Chen SR, Shen YP, Chang CY, Su YC, Chen LC, Wu YT. Long-term outcome after perineural injection with 5% dextrose for carpal tunnel syndrome: a retrospective follow-up study. Rheumatology (Oxford). 2021 Feb 1;60(2):881-887. doi: 10.1093/rheumatology/keaa361. PMID 32856082